CLINICAL TRIAL: NCT04266236
Title: Ultrasound-guided Lumbar Plexus Combined with Quadratus Lumborum Block Using Single-needle Technique with Shamrock Method for Hip Arthroplasty
Brief Title: LPB Combined with QLB Using Single-needle Technique (LPQLB-SNT) for Hip Arthroplasty
Acronym: LPQLB-SNT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaofeng WANG, Attending doctor, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-031
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Hip Osteoarthritis; Anesthesia, Local; Hip Fractures; Osteonecrosis of Femoral Head
Keywords: lumbar plexus block; quadratus lumorum block; total hip arthroplasty; single-needle; shamrock approach
MeSH Terms: conditions — Osteoarthritis, Hip; Hip Fractures; Femur Head Necrosis | interventions — Anesthesia, General; Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- L3 LPB technique (P group) (Active Comparator): ultrasound-guided shamrock approach L3 lumbar plexus block with single-needle technique
  Interventions: Procedure: L3 LPB; Drug: 0.375%ropivacaine 25 ml (Raropin); Procedure: General anesthesia with tracheal intubation
- T12 combined with L3 and L4 LPB technique (TP group) (Active Comparator): ultrasound-guided posterior approach thoracic 12 combined with L3 and L4 lumbar plexus block with mulitple-needle technique
  Interventions: Procedure: L3 LPB; Procedure: L4 LPB; Procedure: T12 block; Drug: 0.375%ropivacaine 40 ml (Raropin); Procedure: General anesthesia with tracheal intubation
- L3 LPB combined with QLB (LPQLB-SNT, PQ group) (Experimental): ultrasound-guided shamrock approach L3 lumbar plexus block combined with quadratus lumborum block with single-needle technique
  Interventions: Procedure: L3 LPB; Procedure: L3 QLB; Drug: 0.375%ropivacaine 40 ml (Raropin); Procedure: General anesthesia with tracheal intubation

INTERVENTIONS:
Procedure: L3 LPB — ultrasound-guided L3 lumbar plexus block
Procedure: L4 LPB — ultrasound-guided L4 lumbar plexus block
  Arms: T12 combined with L3 and L4 LPB technique (TP group)
Procedure: T12 block — ultrasound-guided thoracic 12th segment nerve block
  Arms: T12 combined with L3 and L4 LPB technique (TP group)
Procedure: L3 QLB — ultrasound-guided quadratus lumborum block at L3 level
  Arms: L3 LPB combined with QLB (LPQLB-SNT, PQ group)
Drug: 0.375%ropivacaine 25 ml (Raropin) — 0.375%ropivacaine (Raropin) 25ml will be given
  Arms: L3 LPB technique (P group)
Drug: 0.375%ropivacaine 40 ml (Raropin) — 0.375%ropivacaine (Raropin) 40ml will be given
  Arms: L3 LPB combined with QLB (LPQLB-SNT, PQ group); T12 combined with L3 and L4 LPB technique (TP group)
Procedure: General anesthesia with tracheal intubation — General anesthesia with tracheal intubation will be induced with sufentanil, propofol, vecuronium for every patient before the operation and maintained with sevoflurane during the operation

SUMMARY:
Total hip arthroplasty (THA) is one of the most successful orthopedic procedures to effectively relieve pain and restore function in patients with hip osteoarthritis, osteonecrosis of femoral head and hip fracture.The Lumbar Plexus Block (LPB) is currently used as the standard regional anesthesia technique to provide postoperative pain management after THA. The lumbar plexus (LP) originates from T12 to L5. In general, multiple-needle nerve blockade procedure is needed to block different branches of LP. Therefore, we need more time to finish the regional anethesia procedure and it's not easy for an inexperienced anesthesiologist to master the technique absolutely. In addition, multiple injections will increase the discomfort of the patients. We aim to investigate the effects of lumbar plexus combined with quadratus lumborum block using single-needle technique with Shamrock method as an alternative regional anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) between 18.5 and 30kg/m2 and the weight ≥50kg
2. American Society of Anesthesiologists (ASA) classification I-II
3. Postero-lateral operative incision approach unilateral hip arthroplasty
4. Aged 18-75

Exclusion Criteria:

1. Patient refusal
2. Patients with coagulopathy or on therapeutic anticoagulation
3. Pregnancy
4. Multiple trauma
5. Hypersensitivity or allergy to ropivacaine
6. History of ankylosing spondylitis or spinal surgery
7. Lower extremity neuropathy
8. Unable to communicate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
sensory block assessment | 30 minutes after nerve block procedure
  The sensory block will be assessed by cold alcohol swab and pinprick at lateral, anterior and medial areas of thigh and postero-lateral area of gluteus using a 0 to 2 point scale. 0= no block, patients can feel cold; 1= analgesic block, patient can feel touch but not cold; 2= anesthetic block, patient cannot feel cold or touch.

SECONDARY OUTCOMES:
postoperative static pain at timepoint 1 | at 30mins after the patient recover from general anesthesia
  Visual Analog Scale (VAS) score (0-10, 0 means no pain, 10 means the worst pain) of pain at rest will be recorded at several points of time within 24 hours after surgery: 1) 30mins after the patient recover from general anesthesia in postanesthesia care unit (PACU); 2) 6 hours after surgery;3) 12 hours after surgery; 4) 24 hours after surgery
postoperative static pain at timepoint 2 | at 6 hours after surgery
  Visual Analog Scale (VAS) score (0-10, 0 means no pain, 10 means the worst pain) of pain at rest will be recorded at several points of time within 24 hours after surgery: 1) 30mins after the patient recover from general anesthesia in postanesthesia care unit (PACU); 2) 6 hours after surgery;3) 12 hours after surgery; 4) 24 hours after surgery
postoperative static pain at timepoint 3 | at 12 hours after surgery
  Visual Analog Scale (VAS) score (0-10, 0 means no pain, 10 means the worst pain) of pain at rest will be recorded at several points of time within 24 hours after surgery: 1) 30mins after the patient recover from general anesthesia in postanesthesia care unit (PACU); 2) 6 hours after surgery;3) 12 hours after surgery; 4) 24 hours after surgery
postoperative static pain at timepoint 4 | at 24 hours after surgery
  Visual Analog Scale (VAS) score (0-10, 0 means no pain, 10 means the worst pain) of pain at rest will be recorded at several points of time within 24 hours after surgery: 1) 30mins after the patient recover from general anesthesia in postanesthesia care unit (PACU); 2) 6 hours after surgery;3) 12 hours after surgery; 4) 24 hours after surgery
Performance time of block | During nerve block procedure
  Performance time is defined as the time from insertion of the block needle (skin puncture) until finishing local anaesthetic (LA) injection
intraoperative sufentanil dosage | during the operation
  The total intraoperative sufentanil dosage will be recorded
Incidence of block related adverse events | within 24hours after nerve block procedure
  Intraoperative and postoperative adverse events such as vascular puncture, local anesthetic systemic toxicity, epidural spread, etc.
Cumulative doses of intraoperative vasoactive medications | during the operation
  Cumulative doses of intraoperative vasoactive medications (urapidil, atropine, ephedrine and deoxyepinephrine, etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data with patient identification will not be publicly accessible after the study.

REFERENCES:
- [Derived] Wang X, Zhang J, Xie Z, Chen Y, Yonglin-Chen, Rao Z, Zhang H. Efficacy and safety of combined lumbar plexus and quadratus lumborum block via Shamrock approach at L3 in total hip arthroplasty: a prospective randomized controlled trial. Trials. 2025 Nov 4;26(1):467. doi: 10.1186/s13063-025-09195-w. PMID 41188948
- [Derived] Wang X, Zhang H, Chen Y, Xie Z, Chen M, Chen Y, Zhang J. The anesthetic efficacy of ultrasound-guided lumbar plexus combined with quadratus lumborum block with Shamrock approach in total hip arthroplasty: study protocol for a randomized controlled trial. Trials. 2023 Sep 18;24(1):596. doi: 10.1186/s13063-023-07619-z. PMID 37718446